CLINICAL TRIAL: NCT01670513
Title: A Phase 2 Dose Ranging, Evaluator-Blinded Study to Evaluate the Safety of Topical IDP-118
Acronym: IDP-118
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPSI-IDP-118-P2-01
Record Dates: First submitted 2012-05-31; First posted 2012-08-22 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDP-118 Low Strength (Experimental): IDP-118 Low Strength
  Interventions: Drug: IDP-118 Low Strength
- IDP-118 High Strength (Experimental): IDP-118 High Strength
  Interventions: Drug: IDP-118 High Strength

INTERVENTIONS:
Drug: IDP-118 Low Strength — 8 weeks
  Other Names: IDP-118
  Arms: IDP-118 Low Strength
Drug: IDP-118 High Strength — 8 weeks
  Other Names: IDP-118
  Arms: IDP-118 High Strength

SUMMARY:
Subjects with a clinical diagnosis of plaque psoriasis with 10% to 20% of body surface area affected will be enrolled in the study.

DETAILED DESCRIPTION:
Approximately 60 subjects with a clinical diagnosis of moderate or severe psoriasis (defined as at least of 10 % - 20% treatable Body Surface Area (BSA) and an Investigator's Global Evaluation (IGE) of 3 or 4 at baseline (moderate or severe) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, 18 to 65 (inclusive) years of age.
* Freely given verbal and written informed consent obtained from the subject.
* Clinical diagnosis of psoriasis at the Screening and Baseline visits with
* At least 10% - 20% of total treatable BSA involvement, and
* an Investigator's Global Evaluation score of 3 or 4 ( moderate or severe) on a scale of 0 to 5
* Good general health as determined by the Investigator based on the subject's medical history and physical examination, with Screening hematology, serum chemistry, and urinalysis laboratory values within normal range limits.

Exclusion Criteria:

* Presence of psoriasis that was previously treated with prescription medication prior to the Screening visit and is non-responsive to corticosteroid treatment, as determined by the Investigator.
* Presence of any concurrent skin condition that could interfere with the evaluation of the study drug, as determined by the Investigator.
* History of adrenal disease
* Female who is pregnant, nursing an infant, or planning a pregnancy during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-05 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of HPA axis suppression after treatment with investigational drug product and the comparators | 8 weeks
  To measure the incidence of HPA axis suppression after treatment with investigational drug product and the comparators

SECONDARY OUTCOMES:
To evaluate the safety and cutaneous tolerability of the two formulations and the comparators | 8 weeks
  To evaluate and Local Skin Reactions: Tolerability will be evaluated through assessment of selected local signs and symptoms at the drug-application site: itching, dryness, burning and stinging. In addition the treatment areas will be examined at each visit for significant known drug-related AEs such as skin atrophy, striae, telangiectasia and folliculitis.

OTHER OUTCOMES:
To evaluate efficacy, defined as reduction of severity of disease in a sample target plaque during the course of the study | 8 weeks
  The Investigator will assess the target lesion site affected by psoriasis at each visit. Areas affected by psoriasis (at a minimum 10% BSA) are to be treated with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Todd Plott, MD, Study Director — Medical Monitor
Locations (6):
- United States (6):
  - Dow Clinical Study Site, Santa Rosa, California
  - Dow Clinical Study Site, Clinton Township, Michigan
  - Dow Cliincal Study Site, Fort Gratiot, Michigan
  - Dow Clinical Study Site, Nashville, Tennessee
  - Dow Clinical Study Site, Austin, Texas
  - Dow Clinical Study Site, Norfolk, Virginia